CLINICAL TRIAL: NCT02617316
Title: Analysis of the Different Running Speeds of Strike Patterns: The Efficiency of Shoes
Brief Title: The Different Running Speeds of Strike Patterns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: KMUH-IRB-20130302
Record Dates: First submitted 2015-11-18; First posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: running speeds, strike patterns
MeSH Terms: interventions — Community Health Workers; Shoes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- barefoot first (Other): Ten runners carried on barefoot test first and then in-shoes.
  Interventions: Other: Barefoot; Other: In shoes
- in shoes first (Other): Ten runners carried on in-shoes test first and then barefoot.
  Interventions: Other: Barefoot; Other: In shoes

INTERVENTIONS:
Other: Barefoot — barefoot running test was 20 minutes.
Other: In shoes — In shoes test was 20 minutes.

SUMMARY:
The purpose of this research is to investigate the differences of landing patterns while running in different speed with barefoot and wearing shoe.

DETAILED DESCRIPTION:
Running speed will be adjusted with physical strength and circumstance. When speed changes, whether the landing patterns change or not may be one factor of sports injuries. Therefore, the purpose of this research is to investigate the differences of landing patterns while running in different speed with barefoot and wearing shoe.

ELIGIBILITY:
Inclusion Criteria:

* To jog at least three times a week, each time lasted for more than 20 minutes
* No smokers
* No musculoskeletal diseases within 6 months

Exclusion Criteria:

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The percentage of three kinds of landing patterns. | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lan Y Guo, Ph.D, Study Chair — Department of Sports Medicine, College of Medicine, Kaohsiung Medical University

REFERENCES:
- [Background] Nigg BM, Biomechanics, Load Analysis and Sports Injuries in the Lower-Extremities. Sports Medicine 2(5): 367-379, 1985. Hasegawa H, Yamauchi T, Kraemer WJ. Foot strike patterns of runners at the 15-km point during an elite-level half marathon.Journal Strength Cond Research,21(3): 888-893, 2007. Cavanagh PR, Lafortune MA. Ground reaction forces in distance running. J Biomech 13(5): 397-406, 1980 Shih Y, L KL, TY Shiang. Is the foot striking pattern more important than barefoot or shod conditions in running? Gait Posture 38(3): 490-494, 2013.